CLINICAL TRIAL: NCT02944734
Title: A Multi-center, Randomized, Double-blind, Phase II Clinical Trial to Evaluate the Efficacy and Safety of Combination Therapy vs. Monotherapy of Candesartan and Amlodipine for Dose-Finding in Patients With Essential Hypertension
Brief Title: Comparison of Efficacy and Safety of Combination Therapy and Monotherapy of Candesartan and Amlodipine for Dose-Finding in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SP-AC-002
Record Dates: First submitted 2016-10-24; First posted 2016-10-26 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Essential Hypertension
Keywords: Candesartan; Amlodipine; Hypertension; Vascular Diseases; Cardiovascular Diseases; Antihypertensive Agents; Vasodilator Agents; Angiotensin II Type 1 Receptor Blockers; Angiotensin Receptor Antagonists; Calcium Channel Blockers
MeSH Terms: conditions — Essential Hypertension; Hypertension; Vascular Diseases; Cardiovascular Diseases | interventions — candesartan cilexetil; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (8):
- Candesartan Cilexetil (CC) 8mg (Experimental): Candesartan Cilexetil 8mg, once a day for 8 weeks
  Interventions: Drug: Candesartan Cilexetil 8mg
- CC 16mg (Experimental): Candesartan Cilexetil 16mg, once a day for 8 weeks
  Interventions: Drug: Candesartan Cilexetil 16mg
- Amlodipine(AML) 5mg (Experimental): Amlodipine 5mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 5mg
- AML 10mg (Experimental): Amlodipine 10mg, once a day for 8 weeks
  Interventions: Drug: Amlodipine 10mg
- CC 8mg / AML 5mg (Experimental): Candesartan 8mg and Amlodipine 5mg, once a day for 8 weeks
  Interventions: Drug: Candesartan Cilexetil 8mg; Drug: Amlodipine 5mg
- CC 8mg / AML 10mg (Experimental): Candesartan 8mg and Amlodipine 10mg, once a day for 8 weeks
  Interventions: Drug: Candesartan Cilexetil 8mg; Drug: Amlodipine 10mg
- CC 16mg / AML 5mg (Experimental): Candesartan 16mg and Amlodipine 5mg, once a day for 8 weeks
  Interventions: Drug: Candesartan Cilexetil 16mg; Drug: Amlodipine 5mg
- CC 16mg / AML 10mg (Experimental): Candesartan 16mg and Amlodipine 10mg, once a day for 8 weeks
  Interventions: Drug: Candesartan Cilexetil 16mg; Drug: Amlodipine 10mg

INTERVENTIONS:
Drug: Candesartan Cilexetil 8mg — Candesartan Cilexetil 8mg Daily oral administration for 8 weeks
  Other Names: Atacand 8mg
  Arms: CC 8mg / AML 10mg; CC 8mg / AML 5mg; Candesartan Cilexetil (CC) 8mg
Drug: Candesartan Cilexetil 16mg — Candesartan Cilexetil 16mg Daily oral administration for 8 weeks
  Other Names: Atacand 16mg
  Arms: CC 16mg; CC 16mg / AML 10mg; CC 16mg / AML 5mg
Drug: Amlodipine 5mg — Amlodipine 5mg Daily oral administration for 8 weeks
  Other Names: Norvasc 5mg
  Arms: Amlodipine(AML) 5mg; CC 16mg / AML 5mg; CC 8mg / AML 5mg
Drug: Amlodipine 10mg — Amlodipine 10mg Daily oral administration for 8 weeks
  Other Names: Norvasc 10mg
  Arms: AML 10mg; CC 16mg / AML 10mg; CC 8mg / AML 10mg

SUMMARY:
The purpose of this study is to explore the optimal dose of fixed-dose combination of candesartan cilexetil and amlodipine besylate by examining the safety and efficacy of the combination therapy compared to each of the monotherapy in patients with essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients greater than or equal to 19 years of age
2. Subject who was diagnosed with essential hypertension or after administer the antihypertensive drug (Subject who may temporarily suspend antihypertensive treatment based on doctor's decision)
3. Subject who have voluntarily agreed to participate in the trial and signed the written informed consent form

Exclusion Criteria:

1. Subject with severe hypertension (in a selected arm with msSBP ≥ 200 mmHg or msDBP ≥ 115 mmHg) during the Screening and Randomized Trial.
2. Subject with difference of the blood pressure of over 20 mmHg for SBP or 10 mmHg for diastolic blood pressure (DSP) between three consecutive measurements in a selected arm during the screening visit
3. Secondary hypertension (such as, coarctation of the aorta, primary hyperaldosteronism, renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.)
4. Symptomatic orthostatic hypotension
5. Severe heart failure( New York Heart Association(NYHA) Class III/IV)
6. Subject with acute coronary syndrome(myocardial infarction or unstable angina), peripheral vascular disease within the past 6 months
7. History of switching to another Antiarrhythmic drugs(not including electrolyte correction), or received Cardioversion or ICU treatment within the past 6 months
8. Type 1 diabetes mellitus or Uncontrolled Type 2 diabetes mellitus (HbA1c > 9.0%)
9. Subject with Haemodynamic disturbance, heart valve disease with structural defects
10. Severe cerebrovascular disease (stroke, cerebral infarction, or cerebral hemorrhage, etc. within the past 6 months)
11. Severe eye disease (retinal hemorrhage, visual impairment, retinal microaneurysm, etc. within the past 6 months)
12. Autoimmune diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
13. Chronic inflammatory disease requiring continuous anti-inflammatory treatment
14. Clinically significant Renal or liver impairment, or laboratory abnormalities such as Ccr: below 30ml/min or Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) > 3 x Upper Limit Normal (ULN)
15. Hypokalaemia(Serum potassium < 3.5 mmol/L) or hyperkalaemia(Serum potassium > 5.5 mmol/L)
16. Subject with gastrointestinal disease(such as Crohn's disease, gastric ulcer, acute or chronic pancreatitis) or history of gastrointestinal surgery(not including appendectomy or hernia surgery) that might significantly alter the absorption of the drug
17. history of allergy or hypersensitivity to Angiotensin II Receptor Blockers(Candesartan) or Calcium Channel Blocker(amlodipine)
18. Subject with heredity defects such as galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption
19. Subject requiring concomitant use of other antihypertensive or contraindicated drugs( Tizanidine, dolasetron, Itraconazole, potassium, potassium-sparing diuretics, etc.) during the clinical trial
20. history of malignant tumors within the past 5 years
21. history of alcohol or drug abuse
22. Pregnant women and lactating mothers
23. Women who is planning to be pregnant during or 2 months after the study, or women or men who are not using medically acceptable methods of contraception *

    * progestin oral or implant contraceptive, intra-uterine device, condom, partner with surgical sterilization, etc.
24. Use of other investigational products within the past 1 month
25. Subject who are judged by the investigator unsuitable to participate in the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change mean sitting Diastolic Blood Pressure (msDBP) at week 8 compared to baseline | Week 8

SECONDARY OUTCOMES:
Change mean sitting Diastolic Blood Pressure (msDBP) at week 4 compared to baseline | Week 4
Change mean sitting Systolic Blood Pressure (msSBP) at week 4 and 8 compared to baseline | Week 4 and 8
Proportion of patients achieving treatment goal at week 4 and 8: < 140/90 mmHg | Week 4 and 8
  Joint National Committee VII Guideline Treatment goal: < 140/90 mmHg (< 130/80 mmHg, diabetic or chronic renal failure patient)
Blood Pressure Response rate at week 4 and 8: msSBP reduction ≥ 20 mmHg and msDBP reduction ≥ 10 mmHg | Week 4 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Chong-Jin Kim, Study Director — KyungHee University Hospital at Gangdong
Locations (23):
- South Korea (23):
  - Catholic University of Korea Bucheon St. Mary's Hospital, Wonmi-gu, Bucheon
  - Inje University Busan Paik Hospital, Busanjin-gu, Busan
  - Pusan National University Hospital, Seo-gu, Busan
  - Keimyung University Dongsan Medical Center, Joong-gu, Daegu
  - Kyungpook National University Hospital, Joong-gu, Daegu
  - Daegu Catholic University Medical Center, Nam- Gu, Daegu
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Dongguk University Ilsan Hospital, Ilsandong-gu, Goyang-si, Gyeoggi-do
  - Chonnam National University Hospital, Dong-Gu, Gwangju
  - Catholic University of Korea Uijeongbu St. Mary's hospital, Uijeongbu-si, Gyeoggi-do
  - Gachon University Gil Hospital, Namdong-gu, Incheon
  - St. Carollo General Hospital, Suncheon-si, Jeollanam-do
  - Catholic University of Korea St. Paul's Hospital, Dongdaemun-gu, Seoul
  - KyungHee University Medical Center, Dongdaemun-gu, Seoul
  - Hallym University Kangdong Sacred Heart Hospital, Gangdong-gu, Seoul
  - Kyung Hee University Hospital at Gangdong, Gangdong-Gu, Seoul
  - VHS( Veterans Medical Service) Medical Center, Gangdong-gu, Seoul
  - Konkuk University Medical Center, Gwangjin-gu, Seoul
  - Seoul National University Hospital, Jongro-gu, Seoul
  - Catholic University of Korea Seoul St. Mary's Hospital, Seocho-Gu, Seoul
  - Korea University Anam Hospital, Seongbuk-Gu, Seoul
  - Catholic University of Korea Yeouido St. Mary's Hospital, Yeongdeungpo-gu, Seoul
  - Ulsan University Hospital, Dong-gu, Ulsan

REFERENCES:
- [Derived] Sohn IS, Kim CJ, Ahn T, Youn HJ, Jeon HK, Ihm SH, Cho EJ, Chung WB, Chae SC, Kim WS, Nam CW, Park SM, Choi JY, Kim YK, Hong TJ, Lee HY, Cho JH, Shin ES, Yoon JH, Yang TH, Jeong MH, Lee JH, Park JI. Efficacy and Tolerability of Combination Therapy Versus Monotherapy with Candesartan and/or Amlodipine for Dose Finding in Essential Hypertension: A Phase II Multicenter, Randomized, Double-blind Clinical Trial. Clin Ther. 2017 Aug;39(8):1628-1638. doi: 10.1016/j.clinthera.2017.06.014. Epub 2017 Jul 19. PMID 28734660